CLINICAL TRIAL: NCT03355430
Title: Simultaneous Corneal Wavefront-Guided Trans-PRK and Corneal Collagen Crosslinking After ICRS Implantation for Moderate Keratoconus
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2016-0403
Record Dates: First submitted 2017-11-20; First posted 2017-11-28 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Moderate Keratoconus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- moderate keratoconus group: moderate keratoconus group underwent combined corneal wavefront-guided transepithelial photorefractive keratectomy (tPRK) and accelerated corneal collagen cross-linking (CXL) after intracorneal ring segment (ICRS) implantation
  Interventions: Procedure: combined corneal wavefront-guided transepithelial photorefractive keratectomy (tPRK); Procedure: accelerated corneal collagen cross-linking (CXL)

INTERVENTIONS:
Procedure: combined corneal wavefront-guided transepithelial photorefractive keratectomy (tPRK) — After at least 1 month (average 2.7 ± 1.1 months; range 1 to 4 months), all patients were scheduled for combined corneal wavefront-guided tPRK and accelerated CXL treatment. tPRK between the corneal ring segments was performed using an excimer laser (Amaris 1050 Excimer Laser platform; Schwind eye-tech-solutions GmbH and Co KG, Kleinostheim, Germany).
Procedure: accelerated corneal collagen cross-linking (CXL) — After at least 1 month (average 2.7 ± 1.1 months; range 1 to 4 months), all patients were scheduled for combined corneal wavefront-guided tPRK and accelerated CXL treatment. tPRK between the corneal ring segments was performed using an excimer laser (Amaris 1050 Excimer Laser platform; Schwind eye-tech-solutions GmbH and Co KG, Kleinostheim, Germany).

SUMMARY:
The investigators aim to investigate the effects of combined corneal wavefront-guided transepithelial photorefractive keratectomy (tPRK) and accelerated corneal collagen cross-linking (CXL) after intracorneal ring segment (ICRS) implantation in patients with moderate keratoconus. Medical records of 23 eyes of 23 patients undergoing combined tPRK and CXL after ICRS implantation were retrospectively analyzed. Uncorrected distance visual acuity (UDVA), corrected distance visual acuity (CDVA), manifest refraction spherical equivalent (MRSE), corneal indices based on Scheimpflug tomography, higher-order aberrations (HOAs), and corneal biomechanical properties were evaluated before and after ICRS implantation, and at 1, 3, and 6 months after combined tPRK and CXL. Corneal biomechanical properties were measured using the dynamic Scheimpflug analyzer at approximately the same time of day.

DETAILED DESCRIPTION:
The investigators aim to investigate the effects of combined corneal wavefront-guided transepithelial photorefractive keratectomy (tPRK) and accelerated corneal collagen cross-linking (CXL) after intracorneal ring segment (ICRS) implantation in patients with moderate keratoconus. Medical records of 23 eyes of 23 patients undergoing combined tPRK and CXL after ICRS implantation were retrospectively analyzed. Uncorrected distance visual acuity (UDVA), corrected distance visual acuity (CDVA), manifest refraction spherical equivalent (MRSE), corneal indices based on Scheimpflug tomography, higher-order aberrations (HOAs), and corneal biomechanical properties were evaluated before and after ICRS implantation, and at 1, 3, and 6 months after combined tPRK and CXL. Corneal biomechanical properties were measured using the dynamic Scheimpflug analyzer at approximately the same time of day. The dynamic Scheimpflug analyzer automatically calculated corneal deformation amplitude, radius values, and maximal concave power when the cornea is deformed to its greatest curvature by the air puff. The deformation amplitude is defined as the maximum amplitude when the cornea is deformed to its greatest concave curvature and is influenced by corneal stiffness. The radius values represent the central concave curvature at the highest concavity (depressed to the highest concavity), while maximal concave power is the inverse radius of the curvature at the highest concavity.

ELIGIBILITY:
Inclusion Criteria:

* intolerant to contact lenses
* moderate keratoconus without apical scarring
* if progression had been noted over the previous 6 months
* All included patients underwent combined corneal wavefront-guided tPRK and CXL at least 1 month (average 2.7 ± 1.1 months; range 1 to 4 months) after ICRS implantation.

Exclusion Criteria:

* central or para-central corneal scarring
* central pachymetry < 400 microns
* corneal endothelial cell density of less than 2000 cells/mm2
* systemic autoimmune disease
* a history of herpetic corneal disease
* pregnancy
* lactation
* severe dry eye syndrome

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patient was intolerant to contact lenses, had moderate keratoconus without apical scarring, and if progression had been noted over the previous 6 months. All included patients underwent combined corneal wavefront-guided tPRK and CXL at least 1 month (average 2.7 ± 1.1 months; range 1 to 4 months) after ICRS implantation. We excluded patients with central or para-central corneal scarring, central pachymetry < 400 microns, corneal endothelial cell density of less than 2000 cells/mm2, systemic autoimmune disease, a history of herpetic corneal disease, pregnancy, lactation, or severe dry eye syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2016-07-07 (Actual); Primary Completion 2017-01-02 (Actual); Study Completion 2017-01-02 (Actual)

PRIMARY OUTCOMES:
visual acuity | Pre-operation (baseline)
  visual acuity in eyes undergoing combined corneal wavefront-guided transepithelial photorefractive keratectomy and accelerated corneal collagen cross-linking after intracorneal ring segment implantation in patients with moderate keratoconus
visual acuity | 1 minute before tPRK-CXL(transepithelial photorefractive keratectomy-accelerated corneal collagen cross-linking)
  visual acuity in eyes undergoing combined corneal wavefront-guided transepithelial photorefractive keratectomy and accelerated corneal collagen cross-linking after intracorneal ring segment implantation in patients with moderate keratoconus
visual acuity | 1 month after tPRK-CXL
  visual acuity in eyes undergoing combined corneal wavefront-guided transepithelial photorefractive keratectomy and accelerated corneal collagen cross-linking after intracorneal ring segment implantation in patients with moderate keratoconus
visual acuity | 3-month after tPRK-CXL
  visual acuity in eyes undergoing combined corneal wavefront-guided transepithelial photorefractive keratectomy and accelerated corneal collagen cross-linking after intracorneal ring segment implantation in patients with moderate keratoconus
visual acuity | 6-month after tPRK-CXL
  visual acuity in eyes undergoing combined corneal wavefront-guided transepithelial photorefractive keratectomy and accelerated corneal collagen cross-linking after intracorneal ring segment implantation in patients with moderate keratoconus

SECONDARY OUTCOMES:
Corneal indices | Pre-operation (baseline)
  Multiple corneal indices were measured at the 8-mm zone using the Scheimpflug tomography system (Pentacam HR; OCULUS).
Corneal indices | 1 minute before tPRK-CXL
  Multiple corneal indices were measured at the 8-mm zone using the Scheimpflug tomography system (Pentacam HR; OCULUS).
Corneal indices | 1 month after tPRK-CXL
  Multiple corneal indices were measured at the 8-mm zone using the Scheimpflug tomography system (Pentacam HR; OCULUS).
Corneal indices | 3-month after tPRK-CXL
  Multiple corneal indices were measured at the 8-mm zone using the Scheimpflug tomography system (Pentacam HR; OCULUS).
Corneal indices | 6-month after tPRK-CXL
  Multiple corneal indices were measured at the 8-mm zone using the Scheimpflug tomography system (Pentacam HR; OCULUS).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee H, Kang DSY, Ha BJ, Choi JY, Kim EK, Seo KY, Kim TI. Visual rehabilitation in moderate keratoconus: combined corneal wavefront-guided transepithelial photorefractive keratectomy and high-fluence accelerated corneal collagen cross-linking after intracorneal ring segment implantation. BMC Ophthalmol. 2017 Dec 29;17(1):270. doi: 10.1186/s12886-017-0666-1. PMID 29284455